CLINICAL TRIAL: NCT04164004
Title: Randomized Trial of Patient-Reported Outcome Measurement in Heart Failure Clinic
Brief Title: Patient-Reported Outcome Measurement in Heart Failure Clinic
Acronym: PRO-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Sandhu, Advanced Heart Failure Fellow, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 53713
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Quality of life; Patient-reported outcomes; Quality of care; Implementation research
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Collection of Patient-Reported Health Status (KCCQ-12 Arm) (Experimental): Patients in the KCCQ-12 arm will undergo KCCQ-12 assessment of patient-reported heart failure health status in the electronic health record at each heart failure clinic visit beginning at the start of the trial. Assessment results will be available to clinicians in the electronic health record when making treatment decisions during each clinic visit.
  Interventions: Other: Kansas City Cardiomyopathy Questionnaire-12
- Usual Care (Active Comparator): Patients in the usual care arm will not complete KCCQ-12 assessments in the electronic health record with clinic visits. They will complete a KCCQ-12 assessment at baseline that will not be available to the treating clinician.
  Interventions: Other: Kansas City Cardiomyopathy Questionnaire-12

INTERVENTIONS:
Other: Kansas City Cardiomyopathy Questionnaire-12 — Health status assessment will be completed using the well-validated Kansas City Cardiomyopathy Questionnaire-12 prior to or at the time of heart failure clinic visits.
  Other Names: KCCQ-12

SUMMARY:
This is a randomized study evaluating the effect of routinely collecting a standardized questionnaire of heart failure health status during heart failure clinic visits. Participants will be randomized to early or delayed implementation of a validated health-related quality of life survey (the Kansas City Cardiomyopathy Questionnaire). Participants randomized to early implementation will be given this 12-question survey at each heart failure clinic visit at the beginning of the study; their heart failure clinician will have access to survey results but will continue to manage participants based on standard treatment practice. Patients randomized to delayed implementation will start receiving the survey at each clinic visit one year later. By comparing the health status and treatment rates between early and delayed implementation, this study will determine the impact of standardized health status assessment on patient outcomes and clinician decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Stanford Heart Failure clinic visit during enrollment period

Exclusion Criteria:

* Seen in amyloid clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1249 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Sandhu, MD, MS, Principal Investigator — Instructor of Medicine; Paul A Heidenreich, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Stanford Hospital & Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandhu AT, Calma J, Skye M, Kalwani N, Zheng J, Schirmer J, Din N, Brown Johnson C, Gupta A, Lan R, Yu B, Spertus JA, Heidenreich PA. Clinical Impact of Routine Assessment of Patient-Reported Health Status in Heart Failure Clinic: The PRO-HF Trial. Circulation. 2024 May 28;149(22):1717-1728. doi: 10.1161/CIRCULATIONAHA.124.069624. Epub 2024 Apr 7. PMID 38583147
- [Derived] Brown-Johnson C, Calma J, Amano A, Winget M, Harris SR, Vilendrer S, Asch SM, Heidenreich P, Sandhu AT, Kalwani NM. Evaluating the Implementation of Patient-Reported Outcomes in Heart Failure Clinic: A Qualitative Assessment. Circ Cardiovasc Qual Outcomes. 2023 May;16(5):e009677. doi: 10.1161/CIRCOUTCOMES.122.009677. Epub 2023 Apr 28. PMID 37114990
- [Derived] Sandhu AT, Zheng J, Kalwani NM, Gupta A, Calma J, Skye M, Lan R, Yu B, Spertus JA, Heidenreich PA. Impact of Patient-Reported Outcome Measurement in Heart Failure Clinic on Clinician Health Status Assessment and Patient Experience: A Substudy of the PRO-HF Trial. Circ Heart Fail. 2023 Feb;16(2):e010280. doi: 10.1161/CIRCHEARTFAILURE.122.010280. Epub 2022 Nov 5. PMID 36334312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Routine Collection of Patient-Reported Health Status (KCCQ-12 Arm) | Usual Care
Started | 625 | 624
Completed | 624 | 624
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Collection of Patient-Reported Health Status (KCCQ-12 Arm) | Usual Care | Total
Number analyzed (Participants) | 624 | 624 | 1248
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.1 [52.2 to 73.0] | 63.7 [51.4 to 72.4] | 63.9 [51.8 to 72.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 237 | 485
  Male | 376 | 387 | 763
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 56 | 101
  Not Hispanic or Latino | 551 | 526 | 1077
  Unknown or Not Reported | 28 | 42 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 68 | 75 | 143
  Native Hawaiian or Other Pacific Islander | 6 | 9 | 15
  Black or African American | 30 | 27 | 57
  White | 412 | 398 | 810
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 104 | 112 | 216
Region of Enrollment [Number; unit: participants]
  United States | 624 | 624 | 1248
Heart Failure or Cardiomyopathy Diagnosis [Count of Participants; unit: Participants] | 542 | 547 | 1089
Prior HF Clinic Encounter [Number; unit: participants] | 520 | 526 | 1046

OUTCOME MEASURES:

1. Primary Outcome: Kansas City Cardiomyopathy Questionnaire-12 Score
Description: The first KCCQ-12 score collected one year after randomization will be compared between the KCCQ-12 and usual care arms. KCCQ-12 scores will be collected in the usual care arm starting one year after randomization. Scores will be adjusted for baseline KCCQ-12 in both arms. This will be the primary effectiveness outcome. KCCQ-12 has 4 domains (Physical Limitation Score, Symptom Frequency Score, Quality of Life Score, Social Limitation Score) and one Summary Score. Domain scores are scaled 0-100, and the overall score is the average of the domain scores. For the domain and overall scores, 0 denotes the lowest reportable health status and 100 the highest. Higher values represent a better outcome.
Time Frame: Collected at the first heart failure clinic visit at least one year post-randomization or via telephone interview 15 months post-randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Routine Collection of Patient-Reported Health Status (KCCQ-12 Arm) | Usual Care
Number analyzed (Participants) | 528 | 513
score on a scale | 79.4 (1.0) | 79.7 (1.0)

2. Primary Outcome: Kansas City Cardiomyopathy Questionnaire-12 Response Rate
Description: Frequency of KCCQ-12 response at each clinic visit among patients in the KCCQ-12 arm. This will be the primary implementation outcome. The rate will be calculated as the number of responses divided by the total number of requests to complete the survey.
Time Frame: 1 year
Population: Participants in the KCCQ-12 arm
Measure: Count of Units; unit: Requests
Units Other Than Participants: Requests
Arm/Group | Routine Collection of Patient-Reported Health Status (KCCQ-12 Arm)
Number analyzed (Participants) | 624
Number analyzed (Requests) | 1526
Requests | 1331

3. Secondary Outcome: Percentage of Patients on Beta-blocker Therapy Among Patients With Reduced Ejection Fraction
Description: Beta-blocker therapy use among the sub-group of patients with left ventricular ejection fraction ≤ 40%.
Time Frame: Evaluated at the first heart failure clinic visit at least one year post-randomization or via telephone interview 15 months post-randomization
Reporting Status: Not Posted

4. Secondary Outcome: Median Dose of Beta-Blocker Therapy Among Patients With Reduced Ejection Fraction
Description: Among those patients on beta-blocker therapy, the specific medication and dose will be collected.
Time Frame: as for outcome 3
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Patients on Renin-Angiotensin-Aldosterone System Inhibitors Among Patients With Reduced Ejection Fraction
Description: Use of any renin-angiotensin-aldosterone system inhibitors among the sub-group of patients with left ventricular ejection fraction ≤ 40%. These include angiotensin-converting enzyme inhibitor, angiotensin receptor blockers, or angiotensin receptor-neprilysin inhibitors.
Time Frame: as for outcome 1
Reporting Status: Not Posted

6. Secondary Outcome: Median Dose of Renin-Angiotensin-Aldosterone System Inhibitors Among Patients With Reduced Ejection Fraction
Description: Among those patients on renin-angiotensin-aldosterone system inhibitors with left ventricular ejection fraction ≤ 40%, the specific medication and dose will be collected.
Time Frame: as for outcome 1
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Patients on Mineralocorticoid Receptor Antagonist Among Patients With Reduced Ejection Fraction
Description: Mineralocorticoid receptor antagonist use among the sub-group of patients with left ventricular ejection fraction ≤ 40%.
Time Frame: as for outcome 1
Reporting Status: Not Posted

8. Secondary Outcome: Median Dose of Mineralocorticoid Receptor Antagonist Among Patients With Reduced Ejection Fraction
Description: Among the sub-group of patients with left ventricular ejection fraction ≤ 40% on Mineralocorticoid Receptor Antagonist therapy, the specific medication and dose will be collected.
Time Frame: as for outcome 1
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Patients on Mineralocorticoid Receptor Antagonist Among Patients With Preserved/Mid-Range Ejection Fraction
Description: Mineralocorticoid receptor antagonist use among the sub-group of patients with left ventricular ejection fraction > 40%.
Time Frame: as for outcome 1
Reporting Status: Not Posted

10. Secondary Outcome: Median Dose of Mineralocorticoid Receptor Antagonist Among Patients With Preserved/Mid-Range Ejection Fraction
Description: Among the sub-group of patients with left ventricular ejection fraction > 40% on Mineralocorticoid Receptor Antagonist therapy, the specific medication and dose will be collected.
Time Frame: as for outcome 1
Reporting Status: Not Posted

11. Secondary Outcome: Percentage of Patients on Hydralazine/Nitrate Therapy Among African-American Patients With Reduced Ejection Fraction
Description: Hydralazine/nitrate use among the subgroup of African-American patients with left ventricular ejection fraction ≤ 40%.
Time Frame: as for outcome 1
Reporting Status: Not Posted

12. Secondary Outcome: Median Dose of Hydralazine/Nitrate Therapy Among African-American Patients With Reduced Ejection Fraction
Description: Among the subgroup of African-American patients with left ventricular ejection fraction ≤ 40% on hydralazine/nitrate therapy, the specific dose will be collected
Time Frame: as for outcome 1
Reporting Status: Not Posted

13. Secondary Outcome: Percentage of Patients on Sacubitril-Valsartan Therapy Among the Sub-group of Patients With Reduced Ejection Fraction
Description: Sacubitril-valsartan use among the sub-group of patients with left ventricular ejection fraction ≤ 40%.
Time Frame: as for outcome 1
Reporting Status: Not Posted

14. Secondary Outcome: Median Dose of Sacubitril-Valsartan Therapy Among the Sub-group of Patients With Reduced Ejection Fraction
Description: Among the sub-group of patients with left ventricular ejection fraction ≤ 40% on sacubitril-valsartan, the specific dose will be collected.
Time Frame: as for outcome 1
Reporting Status: Not Posted

15. Secondary Outcome: Percentage of Patients on Sodium/Glucose Cotransporter-2 Inhibitors Therapy Among the Sub-group of Patients With Preserved/Mid-range Ejection Fraction.
Description: Sodium/glucose cotransporter-2 inhibitors use among the sub-group of patients with left ventricular ejection fraction ≤ 40%.
Time Frame: as for outcome 1
Reporting Status: Not Posted

16. Secondary Outcome: Percentage of Patients on Sodium/Glucose Cotransporter-2 Inhibitors Therapy Among the Sub-group of Patients With Left Ventricular Ejection Fraction > 40%.
Description: Sodium/glucose cotransporter-2 inhibitors use among the sub-group of patients with left ventricular ejection fraction > 40%.
Time Frame: as for outcome 1
Reporting Status: Not Posted

17. Secondary Outcome: Percentage of Patients on Ivabradine Therapy Among Patients With Reduced Ejection Fraction With a Heart Rate Above 70 Beats Per Minute on Beta-Blocker Therapy
Description: Ivabradine use among patients with left ventricular ejection fraction ≤ 35% and a heart rate above 70 beats per minute in sinus rhythm.
Time Frame: as for outcome 1
Reporting Status: Not Posted

18. Secondary Outcome: Median Dose of Ivabradine Therapy Among Patients With Reduced Ejection Fraction With a Heart Rate Above 70 Beats Per Minute on Beta-Blocker Therapy
Description: Among patients with left ventricular ejection fraction ≤ 35% and a heart rate above 70 beats per minute in sinus rhythm on ivabradine, the medication dose will be collected.
Time Frame: as for outcome 1
Reporting Status: Not Posted

19. Secondary Outcome: Percentage of Patients With a Implantable Cardiac Defibrillator Among Patients With Reduced Ejection Fraction
Description: Presence of an implantable cardiac defibrillator among the sub-group of patients with left ventricular ejection fraction ≤ 35%.
Time Frame: Evaluated through trial completion (first heart failure clinic visit at least one year post-randomization or via telephone interview 15 months post-randomization)
Reporting Status: Not Posted

20. Secondary Outcome: Percentage of Patients With a Cardiac Resynchronization Therapy Device Among Patients With Reduced Ejection
Description: Presence of cardiac resynchronization therapy among the sub-group of patients with left ventricular ejection fraction ≤ 35% with electrocardiogram findings consistent with a left bundle branch block with QRS width >150ms.
Time Frame: as for outcome 19
Reporting Status: Not Posted

21. Secondary Outcome: Percentage of Patients Given Cardiac Rehabilitation Referral Among Patients With Reduced Ejection Fraction
Description: Referral to cardiac rehabilitation among the subgroup of patients with left ventricular ejection fraction ≤ 35%.
Time Frame: as for outcome 19
Reporting Status: Not Posted

22. Secondary Outcome: Number of Medication Adjustments Per Heart Failure Clinic Visit
Description: The number of medication adjustments made at each heart failure clinic visit. These will include dose changes, new medications, and discontinuation of prior medicines.
Time Frame: Within one year post-randomization
Reporting Status: Not Posted

23. Secondary Outcome: Average Daily Loop Diuretic Dose
Description: The specific loop diuretic and dose will be collected. Diuretic doses will be converted into a standard total daily dose of loop diuretic.
Time Frame: Each clinic visit over one year follow-up and first heart failure clinic visit at least one year after randomization
Reporting Status: Not Posted

24. Secondary Outcome: Count of Hospitalizations Per Patient
Description: Heart failure hospitalizations and non-heart failure hospitalizations in the Stanford healthcare system during the follow-up period.
Time Frame: as for outcome 19
Reporting Status: Not Posted

25. Secondary Outcome: Count of Emergency Department Visits Per Patient
Description: Stanford emergency department visits during the follow-up period.
Time Frame: as for outcome 19
Reporting Status: Not Posted

26. Secondary Outcome: Count of Heart Failure Clinic Visits Per Patient
Description: Stanford heart failure clinic visits during the followup period.
Time Frame: as for outcome 19
Reporting Status: Not Posted

27. Secondary Outcome: Count of Telephone Encounters Per Patient
Description: Stanford heart failure telephone encounters during the follow-up period.
Time Frame: as for outcome 19
Reporting Status: Not Posted

28. Secondary Outcome: Percentage of Patients Who Undergo Formal Advanced Heart Failure Therapy Evaluation
Description: Formal work-up for heart transplant or LVAD (left ventricular assist device) eligibility
Time Frame: Within one year post-randomization
Reporting Status: Not Posted

29. Secondary Outcome: Quality of Patient Clinic Experience
Description: The results from a 10-question survey with ordinal responses regarding patient experience in clinic to a sub-study of all participants enrolled after the first month.
Time Frame: First clinic visit post-randomization within approximately 14 days
Reporting Status: Not Posted

30. Secondary Outcome: Correlation Between Clinician and Patient Perception of Health Status
Description: Patient and clinician perception of health status will be collected. Patient perception is collected via the KCCQ-12 while clinicians will be surveyed regarding health status. We will determine the correlation between patient and clinician perception using an ordinal scale. We will compare correlation across arms.
Time Frame: First clinic visit post-randomization within approximately 14 days
Reporting Status: Not Posted

31. Secondary Outcome: Cardiovascular Diagnostic Test Frequency
Description: Number of diagnostic tests performed between randomization and one year post-randomization. Diagnostic tests include cardiovascular imaging (echocardiography, MRI, cardiac CT, nuclear scan), invasive testing (coronary angiography, right heart catheterization), or ambulatory rhythm monitoring.
Time Frame: Within one year post-randomization
Reporting Status: Not Posted

32. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire-12 Score Among Patients With Heart Failure or Cardiomyopathy
Description: The first KCCQ-12 score collected one year after randomization will be compared between the KCCQ-12 and usual care arms among patients with heart failure or cardiomyopathy The first KCCQ-12 score collected one year after randomization will be compared between the KCCQ-12 and usual care arms. KCCQ-12 scores will be collected in the usual care arm starting one year after randomization. Scores will be adjusted for baseline KCCQ-12 in both arms. This will be the primary effectiveness outcome. KCCQ-12 has 4 domains (Physical Limitation Score, Symptom Frequency Score, Quality of Life Score, Social Limitation Score) and one Summary Score. Scores are scaled 0-100, where 0 denotes the lowest reportable health status and 100 the highest.
Time Frame: Collected at the first heart failure clinic visit at least one year post-randomization or via telephone interview/web questionnaire 15 months post-randomization
Reporting Status: Not Posted

33. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire-12 Score Among Patients With Sub-optimal Health Status at Baseline
Description: The first KCCQ-12 score collected one year after randomization will be compared between the KCCQ-12 and usual care arms among patients with baseline KCCQ <100 at baseline
Time Frame: as for outcome 32
Reporting Status: Not Posted

34. Secondary Outcome: Number of Total Heart Failure Medication Adjustments
Description: The total number of heart failure medication adjustments. Heart failure medications include beta-blockers, renin-angiotensin-aldosterone system inhibitors, mineralocorticoid receptor antagonists, sodium/glucose cotransporter-2 inhibitors, hydralazine/nitrate therapy, ivabradine, or loop diuretics.
Time Frame: Number of medication adjustments from randomization to one year post randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Routine Collection of Patient-Reported Health Status (KCCQ-12 Arm) | Usual Care
All-Cause Mortality (participants affected / at risk) | 23/624 | 21/624
Serious Adverse Events (participants affected / at risk) | 0/624 | 0/624
Other Adverse Events (participants affected / at risk) | 0/624 | 0/624

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT04164004/Prot_SAP_001.pdf